CLINICAL TRIAL: NCT04192136
Title: NAD+ Precursor Supplementation With Exercise Training to Increase Aerobic Capacity in Friedreich's Ataxia
Brief Title: NAD+ and Exercise in FA
Acronym: ExRx in FA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 19-016634; R01HL149722 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Friedreich Ataxia 1
MeSH Terms: conditions — Friedreich Ataxia 1 | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled trial with a 2x2 factorial design testing the effects of an NAD+ precursor (NR) and exercise.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and the investigator team will be blinded as to the group assignment: NR vs Placebo. All collected data (e.g., questionnaires) will be coded, so initial analysis will be conducted without knowledge of the participant's group status.
  While the assignment of participants to the exercise groups will not be blinded to the participant or majority of the study team, a designated blinded technician will perform the follow-up Cardio Pulmonary Exercise Testing. Follow-Up Cardio Pulmonary Exercise Testing will be performed by a dedicated blinded study team member, an exercise technician, who will not know if the participant was assigned to an arm including the exercise intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nicotinamide Riboside (NR) (Experimental): Investigators will use Good Manufacturing Process (GMP)-grade 300 mg capsules of the dietary supplement nicotinamide riboside (ChromaDex, Irvine CA). Investigators dose based on body weight, and monitor for adverse effects (AEs).
  For individuals with weight > 72 kg: 900 mg po qd x 12 wks.
  For individuals with weight > 48 kg and ≤ 72 kg: 600 mg po qd x 12 wks.
  For individuals with weight 24 ≤ 48 kg: 300 mg po qd x 12 wks.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Matched placebo will contain the same excipients without the active supplement and is generally recognized as safe. The placebo will be covered in an identical capsule (NR will be covered in the same capsule). Doses of placebo will match the body weight schema for dosing of NR. Investigators dose based on body weight, and monitor for adverse effects (AEs).
  For individuals with weight > 72 kg: 900 mg po qd x 12 wks.
  For individuals with weight > 48 kg and ≤ 72 kg: 600 mg po qd x 12 wks.
  For individuals with weight 24 ≤ 48 kg: 300 mg po qd x 12 wks.
  Interventions: Dietary Supplement: Placebo
- Exercise Intervention and NR (Experimental): The exercise program consists of at-home training sessions: 3 aerobic sessions per week on the in-home bike trainer, and 2 resistance exercise sessions per week using resistance bands. All sessions will begin with stretching and brief aerobic warm-up exercise on the in-home bike trainer. On resistance training days, subjects will be given instructions to complete circuits of resistance exercises.
  Participants in this arm will receive both the Exercise Intervention and the NR.
  Interventions: Dietary Supplement: Nicotinamide Riboside; Other: Exercise Intervention
- Exercise Intervention and Placebo (Experimental): The exercise program consists of at-home training sessions: 3 aerobic sessions per week on the in-home bike trainer, and 2 resistance exercise sessions per week using resistance bands. All sessions will begin with stretching and brief aerobic warm-up exercise on the in-home bike trainer. On resistance training days, subjects will be given instructions to complete circuits of resistance exercises.
  Participants in this arm will receive both the Exercise Intervention and the Placebo.
  Interventions: Dietary Supplement: Placebo; Other: Exercise Intervention

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Investigators will use (Good Manufacturing Process) GMP-grade 300 mg capsules of the dietary supplement nicotinamide riboside (ChromaDex, Irvine CA).
  NR is distributed by ChromaDex, Inc., Irvine, CA. NR is available as 300 mg capsules.
  The dietary supplement will be re-labeled by the Hospital of the University of Pennsylvania (HUP) Investigational Drug Service according to FDA regulations, including subject and physician name and NR or Placebo 300 mg capsules.
  Arms: Exercise Intervention and NR; Nicotinamide Riboside (NR)
Dietary Supplement: Placebo — The matched placebo will contain the same excipients without the active supplement and is generally recognized as safe. The placebo will be covered in an identical capsule (NR will be covered in the same capsule).
  Arms: Exercise Intervention and Placebo; Placebo
Other: Exercise Intervention — The exercise program consists of at-home training sessions: 3 aerobic sessions per week on the in-home bike trainer, and 2 resistance exercise sessions per week using resistance bands.
  On aerobic training days, subjects will be given instruction on a recumbent Catrike trainer, titrated such that they spend 20 minutes at their target heart rate as determined by baseline Exercise Stress Test (EST) (60-80% of their heart rate at peak VO2) and as measured by their wearable device.
  On resistance training days, subjects will be given instructions to complete circuits of resistance exercises. Resistance training intensity (as determined by graded resistance bands) will be maintained at 60% of pre-training maximal voluntary contraction for each muscle group.
  Arms: Exercise Intervention and NR; Exercise Intervention and Placebo

SUMMARY:
Randomized, placebo-controlled trial with a 2x2 factorial design testing the effects of an NAD+ precursor (NR) and exercise on VO2max and Si in Friedreich's Ataxia (FA).

The primary objective of this research is to measure the effect of combination administration (NR + exercise) on aerobic capacity (VO2max) in FA. A key secondary objective is to measure the effect of combination administration (NR + exercise) on glucose homeostasis (Si) in FA.

DETAILED DESCRIPTION:
Friedreich's Ataxia (FA) is a progressive neurodegenerative disease affecting 1 in 50,000 individuals in the U.S. Currently, there is no approved treatment.

There is a critical knowledge gap regarding the best ways to intervene to increase aerobic capacity (VO2max on exercise testing) in FA. Exercise is the most potent known stimulus for increasing muscle mass and mitochondrial oxidative phosphorylation (OXPHOS) capacity, increasing VO2max, and increasing insulin sensitivity (Si), however, it has not been studied in FA. One adaptation seen in exercised muscles is an increase in muscle nicotinamide adenine dinucleotide (NAD+), a cofactor required for glycolytic and mitochondrial adenosine triphosphate (ATP) production. In skeletal- and cardiac muscle-specific frataxin (FXN) knock-out animals, NAD+ precursors rescued cardiac function to near-normal, additionally highlighting its translational potential in FA. Nicotinamide riboside (NR) is a NAD+ precursor currently available as a dietary supplement (Tru Niagen ®, ChromaDex, Irvine CA) that is expected to be safe and well-tolerated in adults and children. The central hypothesis is that exercise + NR will increase skeletal muscle mitochondrial OXPHOS and increase muscle mass to increase VO2max in FA. The investigators expect that exercise + NR will also increase Si in this cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Molecular diagnosis of Friedrich's Ataxia (FA).
2. Males and Females, Age 10 to 40 years (inclusive).
3. Girls, 11 years of age and older, must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
4. Not currently meeting exercise guidelines as outlined by The Physical Activity Guidelines for Americans.

   * Children and Adolescents should do 60 minutes (1 hour) or more of moderate-to-vigorous physical activity daily.
   * As a part of their physical activity, children and adolescents should include muscle-strengthening physical activity on at least 3 days a week.
   * Adults should do at least 150 minutes (2 hours and 30 minutes) to 300 minutes (5 hours) a week of moderate-intensity, or 75 minutes (1 hour and 15 minutes) to 150 minutes (2 hours and 30 minutes) a week of vigorous-intensity aerobic physical activity.
   * Adults should also do muscle-strengthening activities of moderate or greater intensity that involve all major muscle groups on 2 or more days a week.
5. Cardiac echocardiogram or cardiac MRI, performed within 1 year of enrollment, showing an LVEF > 45%
6. ECG, performed within 1 year of enrollment, without clinically significant arrhythmia.
7. Weight > 24 kg
8. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Known sensitivity to NR.
2. Concurrent use of any medications, including statins, likely to increase risk of NR toxicity.
3. HgbA1c > 8.5% and/or Diabetes Mellitus (DM) requiring insulin or insulin secretagogue.
4. Use of supraphysiologic steroids.
5. Laboratory abnormalities that indicate clinically significant anemia or bleeding risk. (Hemoglobin < 10 g/dL or Platelets < 100K)
6. Laboratory abnormalities that indicate clinically significant kidney disease using serum creatinine and Modification of Diet in Renal Disease (MDRD) equation. (Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73 m2)
7. Laboratory abnormalities that indicate clinically significant liver disease. (Aspartate Aminotransferase (AST)/Serum Glutamic Oxaloacetic Transaminase (SGOT) 3.0 x Upper Limit of Normal and/or Alanine Aminotransferase (ALT)/Serum Glutamic Pyruvic Transaminase (SGPT) 3.0 x Upper Limit of Normal)
8. Uncontrolled and persistent arrhythmias that are felt to be clinically significant.
9. Known history of moderate or severe left ventricular systolic dysfunction (Left Ventricular Ejection Fraction (LVEF) < 45%)
10. Standard contraindications to exercise testing.
11. Inability to sit and pedal unassisted in a cycle ergometry chair, at a cadence of at least 55 rotations per minute (rpm) during unloaded warm up, in a cycle ergometry chair and complete a maximal Cardio Pulmonary Exercise Test (CPET)
12. Inability to sit and pedal unassisted in a recumbent tricycle.
13. Any contraindication to MRI. Including:

    * Any intra-luminal implant, filter, stent or valve replacement
    * Any type of life assist device, pump, or prosthetic
    * Any vascular clip or clamp
    * Any surgically placed clips or clamps or bands on visceral organs
    * Any intracranial implants of any type other than dental fillings
    * Any non-removable piercings, jewelry, or medicinal patch
    * Any personal history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic examination.
    * Any personal history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation.
    * Inability to lie flat in the MRI scanner for 60-90 minutes.

      * participants who cannot complete the MRI will not be excluded from participation in the remainder of the study procedures if they meet those inclusion and exclusion criteria
14. Use of any investigational agent within 4 weeks of enrollment, except open-label extension phase.
15. Females: pregnant, lactating, or planning to become pregnant during their participation.
16. Any medical condition, in the opinion of the investigator that will interfere with the safe completion of the study.
17. Parents/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Within-Participant Change in V02 Max (Maximal Oxygen Uptake on Cardiopulmonary Exercise Testing) | Baseline to 12 Weeks
  V02 Max will be assessed by completion of an incremental symptom-limited cardio-pulmonary Exercise Stress Test (EST) on a recumbent leg cycle ergometer.

SECONDARY OUTCOMES:
Within-Participant Change in Whole Body Insulin Sensitivity (Si) | Baseline to 12 Weeks
  Whole Body Insulin Sensitivity (Si) will be assessed by completion of a stable isotope tracer-enhanced Oral Glucose Tolerance Test (OGTT). Samples will be collected at 10 time points for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States